CLINICAL TRIAL: NCT01753141
Title: Smoking Treatment and Anxiety Management Program
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH076629-01A1 (NIH)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Nicotine Dependence
Keywords: Cognitive Behavioral Therapy; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Cognitive Behavioral Therapy for smoking cessation plus anxiety sensitivity reduction.
  Interventions: Behavioral: Cognitive Behavioral Therapy for smoking cessation and anxiety sensitivity reduction.
- Control (Active Comparator): Cognitive Behavioral Therapy for smoking cessation.
  Interventions: Behavioral: Cognitive Behavioral Therapy for smoking cessation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for smoking cessation
  Arms: Control
Behavioral: Cognitive Behavioral Therapy for smoking cessation and anxiety sensitivity reduction. — Includes anxiety sensitivity (AS) psychoeducation and interoceptive exposure exercises in addition to regular smoking cognitive behavioral therapy.
  Arms: Active

SUMMARY:
The Smoking Treatment and Anxiety Management Program (STAMP) is a treatment program focused on helping people manage their anxiety while quitting smoking. The study involves coming in to our clinic for 4 treatment sessions, with follow-ups for up to 2 years (a week 1, week 2, month 1, month 3, month 6, year 1, and year 2 follow-up). Participants will be paid $142.50 for their full participation as well as receive 6 weeks of free nicotine replacement patches.

ELIGIBILITY:
Inclusion Criteria:

* Anxiety Sensitivity Index greater than 15
* Daily smoker for at least 1 year
* Less than 45 years old
* Currently smoke at least 8 cigarettes per day
* Report a motivation to quit smoking

Exclusion Criteria:

* History of panic disorder
* Psychotropic medication use (if not stable for 3 months)
* History of significant medical condition
* Current use of smoking cessation pharmacology
* Use of other tobacco products
* Planning to move in the next 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 378 (Actual)
Dates: Start 2008-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index | up to 2 years
  The ASI is a 16-item self-report measure that assesses the fear of consequences of bodily sensations associated with anxiety. Items are rated on a five-point Likert-type scale ranging from 0 (very little) to 4 (very much) and a total score is computed by summing all items. The ASI is hierarchical in structure with one higher order factor (AS) and three subfactors (physical, cognitive, and social concerns). The physical concerns subscale includes items related to the fear of consequences or presence of specific physical sensations (e.g. "When I notice that my heart is beating rapidly, I worry that I might have a heart attack"). The cognitive concerns subscale includes items related to potential mental health implications of sensations (e.g. "When I cannot keep my mind on a task, I worry that I might be going crazy"). The social concerns subscale includes items related to the potential social consequences of physical sensations (e.g. "It is important to me not to appear nervous").

SECONDARY OUTCOMES:
Smoking Status | week 1, week 2, month 1, month 3, month 6, year 1, and year 2 follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States

REFERENCES:
- [Result] Brandt CP, Johnson KA, Schmidt NB, Zvolensky MJ. Main and interactive effects of emotion dysregulation and breath-holding duration in relation to panic-relevant fear and expectancies about anxiety-related sensations among adult daily smokers. J Anxiety Disord. 2012 Jan;26(1):173-81. doi: 10.1016/j.janxdis.2011.10.007. Epub 2011 Nov 6. PMID 22119451
- [Result] Buckner JD, Zvolensky MJ, Schmidt NB. Cannabis-related impairment and social anxiety: the roles of gender and cannabis use motives. Addict Behav. 2012 Nov;37(11):1294-7. doi: 10.1016/j.addbeh.2012.06.013. Epub 2012 Jun 22. PMID 22766487
- [Result] Buckner JD, Joiner TE Jr, Schmidt NB, Zvolensky MJ. Daily marijuana use and suicidality: the unique impact of social anxiety. Addict Behav. 2012 Apr;37(4):387-92. doi: 10.1016/j.addbeh.2011.11.019. Epub 2011 Nov 25. PMID 22154236
- [Result] Capron DW, Blumenthal H, Medley AN, Lewis S, Feldner MT, Zvolensky MJ, Schmidt NB. Anxiety sensitivity cognitive concerns predict suicidality among smokers. J Affect Disord. 2012 May;138(3):239-46. doi: 10.1016/j.jad.2012.01.048. Epub 2012 Feb 26. PMID 22370063
- [Result] Johnson KA, Farris SG, Schmidt NB, Zvolensky MJ. Anxiety sensitivity and cognitive-based smoking processes: testing the mediating role of emotion dysregulation among treatment-seeking daily smokers. J Addict Dis. 2012;31(2):143-57. doi: 10.1080/10550887.2012.665695. PMID 22540436
- [Result] Peasley-Miklus CE, McLeish AC, Schmidt NB, Zvolensky MJ. An examination of smoking outcome expectancies, smoking motives and trait worry in a sample of treatment-seeking smokers. Addict Behav. 2012 Apr;37(4):407-13. doi: 10.1016/j.addbeh.2011.11.037. Epub 2011 Dec 3. PMID 22209026
- [Result] Funk, A. P., Zvolensky, M. J., & Schmidt, N. B. Homework compliance in a brief cognitive-behavioral and pharmacological intervention for smoking. Journal of Smoking Cessation (6): 99-111, 2011.
- [Result] Leventhal AM, Zvolensky MJ, Schmidt NB. Smoking-related correlates of depressive symptom dimensions in treatment-seeking smokers. Nicotine Tob Res. 2011 Aug;13(8):668-76. doi: 10.1093/ntr/ntr056. Epub 2011 Apr 6. PMID 21471305
- [Derived] Rogers AH, Bakhshaie J, Garey L, Piasecki TM, Gallagher MW, Schmidt NB, Zvolensky MJ. Individual differences in emotion dysregulation and trajectory of withdrawal symptoms during a quit attempt among treatment-seeking smokers. Behav Res Ther. 2019 Apr;115:4-11. doi: 10.1016/j.brat.2018.10.007. Epub 2018 Oct 19. PMID 30384961
- [Derived] Zvolensky MJ, Garey L, Allan NP, Farris SG, Raines AM, Smits JAJ, Kauffman BY, Manning K, Schmidt NB. Effects of anxiety sensitivity reduction on smoking abstinence: An analysis from a panic prevention program. J Consult Clin Psychol. 2018 May;86(5):474-485. doi: 10.1037/ccp0000288. PMID 29683703